CLINICAL TRIAL: NCT06546423
Title: Phase I Study of the Infectivity, Safety and Immunogenicity of Two Recombinant, Live-Attenuated, Bovine/Human, Parainfluenza Virus Type 3 (B/HPIV3) Vectored Vaccines Expressing the Fusion Glycoprotein of Human Metapneumovirus (HMPV), Delivered by Nasal Spray to HPIV3-Seropositive Children 24 to <60 Months of Age
Brief Title: Study of the Infectivity, Safety and Immunogenicity of Two Recombinant, Live-Attenuated, B/HPIV3 Vectored Vaccines Expressing the Fusion Glycoprotein of HMPV Delivered by Nasal Spray to HPIV3-Seropositive Children 24 to <60 Months of Age
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other); Vanderbilt University Medical Center (Other); University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR363
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Human Metapneumovirus; Human Parainfluenza Virus Type 3
MeSH Terms: interventions — Ringer's Lactate; Injections

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive B/HPIV3/HMPV-PreF-A vaccine, B/HPIV3/HMPV-F-B365 vaccine or placebo in a 2:2:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To ensure the unbiased clinical evaluation of subjects, all participants' parents/guardians and all staff involved in clinical assessment will remain blinded through completion. To assess the magnitude and duration of vaccine virus replication and ensure continued suitability of these vaccines for this population in this Phase 1 trial, a Scientific Investigator who is not involved in clinical assessment of trial participants, will be unblinded once the final participant in each randomization block has completed the assessment phase on Day 28. Should any concerns arise from this review, these will be shared in a blinded fashion with the Medical Monitor and Sponsor Clinical Safety Office for guidance and assistance. Additionally, this information will be reviewed unblinded by the DSMB in collaboration with the Scientific Investigator and any involved non-study-team consultants before any additional dosing or enrollments proceed.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- B/HPIV3/HMPV-PreF-A vaccine (Active Comparator): A single dose of intranasal B/HPIV3/HMPV-PreF-A will be administered by a Vax300 VaxINator atomization device.
  Interventions: Biological: B/HPIV3/HMPV-PreF-A vaccine
- B/HPIV3/HMPV-F-B365 vaccine (Active Comparator): A single dose of intranasal B/HPIV3/HMPV-F-B365 will be administered by a Vax300 VaxINator atomization device.
  Interventions: Biological: B/HPIV3/HMPV-F-B365 vaccine
- Placebo (Placebo Comparator): A single dose of intranasal Lactated Ringer's Solution for Injection will be administered by a Vax300 VaxINator atomization device.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: B/HPIV3/HMPV-PreF-A vaccine — B/HPIV3/HMPV-PreF-A is a live-attenuated vaccine candidate. The B/HPIV3/HMPV-PreF-A vaccine is provided in a sterile 2.0-mL cryovial, each containing 0.6 mL of vaccine with a titer of approximately 10^6.7 PFU/mL. The vaccine virus concentrate is diluted with Lactated Ringer's Solution for Injection to a dose of approximately 10^5.6 PFU in a 0.2 mL volume.
  Arms: B/HPIV3/HMPV-PreF-A vaccine
Biological: B/HPIV3/HMPV-F-B365 vaccine — B/HPIV3/HMPV-F-B365 is a live-attenuated vaccine candidate. The B/HPIV3/HMPV-F-B365 vaccine is provided in a sterile 2.0-mL cryovial, each containing 0.6 mL of vaccine with a titer of approximately 10^6.3 PFU/mL. The vaccine virus concentrate is diluted with Lactated Ringer's Solution for Injection to a dose of approximately 10^5.6 PFU in a 0.2 mL volume.
  Arms: B/HPIV3/HMPV-F-B365 vaccine
Drug: Placebo — Lactated Ringer's Injection, USP is a sterile, nonpyrogenic solution for fluid and electrolyte replenishment. It will be drawn up in a sterile syringe to a volume of 0.2 mL.
  Other Names: Lactated Ringer's Solution for Injection
  Arms: Placebo

SUMMARY:
HPIV3 and HMPV are viruses that can cause breathing problems in children. The goal of this clinical trial is to look at the safety of 2 experimental HPIV3/HMPV vaccines in HPIV3-seropositive children ≥ 24 months to < 60 months of age. Children will receive B/HPIV3/HMPV-PreF-A vaccine, B/HPIV3/HMPV-F-B365 vaccine, or placebo, and participants will not know which study product they have received.

The main goals of the study are to find out whether these vaccines are well-tolerated and infectious in HPIV3-seropositive children.

The general procedures include daily temperature measurements and daily contact with the participant for the first 28 days, giving a single dose of one of the 2 study vaccines or placebo delivered by nasal sprayer, about 9 in-person visits, a physical examination, 7 clinical assessments, 2 blood samples, 9 nasal swabs and monthly contacts with the participant between Days 29-180.

Additional visits may occur if the child has a respiratory illness, fever, or ear infections. The illness visit will include a nasal swab and a clinical assessment.

DETAILED DESCRIPTION:
This is a blinded, randomized, placebo-controlled study design will be used to evaluate the safety and immunogenicity of the study product in HPIV3-seropositive participants. The study will be performed in approximately 25 HPIV3-seropositive children ≥ 24 months to < 60 months of age. Subjects will be block randomized to receive a single dose of 10^5.6 PFU of B/HPIV3/HMPV-PreF-A, 10^5.6 PFU of B/HPIV3/HMPV-F-B365, or placebo in a 2:2:1 ratio. Enrollment will be continuous unless stopping rules are met or other safety concerns occur. During the enrollment period, the Data and Safety Monitoring Board (DSMB) will perform unblinded safety reviews. After completion of the Day 28 visit of the last participant, an unblinded review of all participants will be performed by the DSMB.

The first 28 days after inoculation are considered the Acute Phase of the study, and the participants' parents/guardians will be contacted daily during the Acute Phase. These contacts will consist either of an in-person evaluation of interim medical history, clinical assessment, and nasal swab, or an interim medical history conducted by a mutually agreed upon communication method. If a child develops a respiratory or febrile illness or otitis media during the acute phase, an in-person evaluation will be performed. During the Acute Phase, the participants will be evaluated for adverse events (AEs) or serious adverse events (SAEs). Between Days 29 and 180 parents/guardians will be asked to contact study staff to report Medically Attended Adverse Events (MAAEs), which will be reported per protocol. Between days 29-180, study staff will contact the participants' parents/guardians monthly and on Day 180 (±7 days) after inoculation to capture any previously unreported MAAEs.

Clinical assessments will be completed and nasal swabs will be obtained on study Days 0, 3, 4, 5, 6, 7, 10, 14 and 28 and whenever febrile or respiratory illnesses or otitis media (solicited AEs) are reported during the first 28 days following inoculation. The nasal swab will be tested for vaccine virus, for respiratory pathogens that are considered adventitious agents, including wild-type HPIV3 and HMPV, and for mucosal IgG and IgA antibody as listed in the schedule of events.

ELIGIBILITY:
Inclusion Criteria:

* ≥24 months of age and <60 months of age at the time of inoculation
* HAI Screening for HPIV3-neutralizing antibody is obtained within the calendar year of inoculation
* Seropositive for HPIV3 antibody, defined as serum HPIV3 HAI titer >1:8
* Pre-inoculation serum sample for HPIV3-neutralizing antibody specimen is obtained no more than 42 days prior to inoculation
* In good health based on review of the medical record, history, and physical examination at the time of inoculation
* Received routine immunizations appropriate for age based on the Advisory Committee on Immunization Practices (ACIP) Recommended Immunization Schedule for Children and Adolescents Aged 18 Years or Younger
* Growing normally for age as demonstrated on a World Health Organization (WHO) growth chart, AND has a current height and weight above the 3rd percentile for age
* Expected to be available for the duration of the study
* Parent/guardian is willing and able to provide written informed consent

Exclusion Criteria:

* <24 months of age and >60 months of age at the time of inoculation.
* Born at less than 34 weeks gestation
* Maternal history of a positive HIV test before or during pregnancy.
* Evidence of chronic disease
* Known or suspected infection or impairment of immunological functions
* Bone marrow/solid organ transplant recipient
* Major congenital malformations, including congenital cleft palate or cytogenetic abnormalities
* Suspected or documented developmental disorder, delay, or other developmental problem
* Cardiac abnormality requiring treatment
* Lung disease or reactive airway disease
* More than one episode of medically diagnosed wheezing in the first year of life
* Wheezing episode or received bronchodilator therapy or racemic epinephrine within the past 12 months
* Wheezing episode or received bronchodilator therapy after the age of 12 months
* Previous receipt of supplemental oxygen therapy in a home setting
* Previous receipt of an investigational HPIV3 or HMPV vaccine
* Previous receipt or planned administration of human immunoglobulin within the past 6 months. Receipt of licensed monoclonal antibody products for passive prophylaxis against RSV (e.g., nirsevimab) within the past 6 months is not a cause for exclusion
* Previous receipt of any blood products within the past 6 months.
* Previous anaphylactic reaction
* Previous vaccine-associated adverse reaction that was Grade 3 or above.
* Known hypersensitivity to any study product component
* Member of a household that contains an infant who is less than 12 months of age at the date of inoculation through the 10th day after inoculation
* Member of a household that, at the date of inoculation through the 10th day after inoculation, contains an immunocompromised individual including but not limited to:

  * a person who is HIV-infected
  * a person who has cancer and has received chemotherapy within the 12 months prior to enrollment
  * a person living with a solid organ or bone marrow transplant
* Attends a daycare facility that does not separate children by age and contains a child <12 months of age at the date of inoculation through the 10th day after inoculation
* Receipt of any of the following prior to enrollment:

  * inactivated influenza vaccine within 3 days prior, or
  * any other inactivated vaccine, messenger RNA (mRNA) vaccine, or live-attenuated rotavirus vaccine within the 14 days prior, or
  * any live vaccine, other than rotavirus vaccine, within the 28 days prior, or
  * another investigational vaccine or investigational drug within 28 days prior, or
  * salicylate (aspirin) or salicylate-containing products within the past 28 days
* Scheduled administration of any of the following after planned inoculation:

  * inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days after, or
  * any live vaccine other than rotavirus within the 28 days after, or
  * any salicylate or salicylate-containing products within the 28 days after, or
  * another investigational vaccine or investigational drug in the 56 days after
* Receipt of any of the following medications within 3 days prior to study enrollment:

  * systemic antibacterial, antiviral, antifungal, anti-parasitic, or antituberculous agents, whether for treatment or prophylaxis, or
  * intranasal medications, or
  * other prescription medications except the permitted concomitant medications listed below
  * Permitted concomitant medications (prescription or non-prescription) include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including (but not limited to) cutaneous (topical) steroids, topical antibiotics, and topical antifungal agents
* Any of the following events at the time of enrollment:

  * fever (temporal or rectal temperature of ≥100.4°F), or
  * upper respiratory signs or symptoms (rhinorrhea, cough, or pharyngitis), or
  * nasal congestion significant enough to interfere with successful inoculation, or
  * otitis media, or
  * contact with a person diagnosed with COVID-19 disease or active SARS-CoV-2 infection within the preceding 10 days

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of Grade 1 or higher solicited AEs; any lower respiratory infections | Day 0 through Day 28
Percentages of vaccinees with a ≥4-fold rise in HPIV3 neutralizing serum antibody titers | Day 28
Percentages of vaccinees with a ≥4-fold rise in HMPV-neutralizing serum antibody titers | Day 28
Peak titers of vaccine virus shed | Study Days 0-28
Proportion of vaccinees shedding of vaccine virus | Day 28
  Detected by immunoplaque assay and/or RT-qPCR, and/or ≥4 fold rise in HPIV3 or HMPV-specific serum antibodies, detected by neutralizing antibody assay or ELISA

SECONDARY OUTCOMES:
Number of MAAEs and SAEs | Day 0 through Day 180
  MAAEs and SAEs from Day 0 through Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Karron, M.D., Principal Investigator — Center for Immunization Research, JHBSPH
Locations (4):
- United States (4):
  - CIR - Rangos, Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - CIR South, Columbia, Maryland
  - University of Rochester Medical Center, Rochester, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to IPD that underlie results in a publication. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants.
Time Frame: After publication
Access Criteria: Qualified researchers